CLINICAL TRIAL: NCT06727058
Title: A Phase 1/2, Randomized, Modified Double-blind, Placebo-controlled, Multi-center, Dose Escalating Study to Evaluate the Safety and Immunogenicity of a Pandemic Flu H5 mRNA Vaccine in Healthy Adults Aged 18 Years and Older
Brief Title: Study to Evaluate Safety and Immunogenicity of a Pandemic Flu H5 mRNA Vaccine in Healthy Adults Aged 18 Years and Older
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: VBS00001; U1111-1309-8833 (Other: WHO ICTRP)
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Influenza Immunization
Keywords: pandemic influenza infection; H5 strain
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Modified double blind (participants; sites, except for those preparing/administering study intervention; and Sponsor will be blinded). Sponsor's internal safety monitoring team will be unblinded if necessary. "Evaluation of the Safety of the sentinel cohorts will be unmasked for the Sponsor's safety Team".
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Low Dose Pandemic flu H5 mRNA vaccine (Experimental): Participants will receive 2 injections of pandemic flu H5 mRNA vaccine 21 days apart (at Day 01 and Day 22)
  Interventions: Biological: Pandemic flu H5 mRNA vaccine
- Group 2: Medium Dose Pandemic flu H5 mRNA vaccine (Experimental): Participants will receive 2 injections of pandemic flu H5 mRNA vaccine 21 days apart (at Day 01 and Day 22)
  Interventions: Biological: Pandemic flu H5 mRNA vaccine
- Group 3: High Dose Pandemic flu H5 mRNA vaccine (Experimental): Participants will receive 2 injections of pandemic flu H5 mRNA vaccine 21 days apart (at Day 01 and Day 22)
  Interventions: Biological: Pandemic flu H5 mRNA vaccine
- Group 4: Placebo (Placebo Comparator): Participants will receive 2 injections of placebo 21 days apart (at Day 01 and Day 22)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Pandemic flu H5 mRNA vaccine — Pharmaceutical Form: Suspension for injection
  Route of Administration: Intramuscular (IM)
  Arms: Group 1: Low Dose Pandemic flu H5 mRNA vaccine; Group 2: Medium Dose Pandemic flu H5 mRNA vaccine; Group 3: High Dose Pandemic flu H5 mRNA vaccine
Other: Placebo — Pharmaceutical Form: Liquid solution for injection
  Route of Administration: Intramuscular (IM)
  Arms: Group 4: Placebo

SUMMARY:
The purpose of this study is to evaluate a pandemic flu H5 strain messenger ribonucleic acid (mRNA) vaccine at 3 dose levels (low, medium, and high) in comparison with placebo in 276 healthy adult participants to select the adequate dose for further clinical development.

The duration per participant will be approximately 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older on the day of inclusion.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile.

OR

• Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to each study intervention administration until at least 12 weeks after the last study intervention administration.

* A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 8 hours before the first dose of study intervention.

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the study intervention components (eg, polyethylene glycol, polysorbate); history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances; any allergic reaction (eg, anaphylaxis) after administration of an mRNA vaccine .
* Previous history of myocarditis, pericarditis, and/or myopericarditis.
* Known history of previous episodes of Guillain-Barré Syndrome (GBS), neuritis (including Bell's palsy), convulsions , encephalitis, transverse myelitis, and vasculitis.
* Participants with an electrocardiogram that is consistent with possible myocarditis or pericarditis or, in the opinion of the investigator, demonstrates clinically relevant abnormalities that may affect participant safety or study results.
* Self-reported thrombocytopenia, contraindicating IM injection based on investigator's judgment.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM injection based on investigator's judgment.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness / infection (according to investigator's judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Alcohol, prescription drug, or substance abuse that, in the opinion of the investigator, might interfere with the study conduct or completion.
* Participant who had acute infectious symptoms or a positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) reverse transcriptase polymerase chain reaction (RT PCR) or antigen test in the past 10 days prior to the first visit (V)01.
* Receipt of any vaccine other than an mRNA vaccine in the 4 weeks preceding study intervention administration or planned receipt of any vaccine other than an mRNA vaccine in the 3 weeks following the second dose of the study intervention .
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Receipt of any mRNA vaccine/product in the 2 months preceding study intervention administration or planned receipt of any mRNA vaccine in the 2 months after the second dose of the study intervention.
* Participation at the time of study enrollment (or in the 4 weeks preceding study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Previous history of participation in an H5 influenza A vaccine study. This includes any influenza subtypes that contain H5 such as H5N1, H5N8, or H5N6.

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Presence of immediate adverse events (AEs) within 30 minutes after each/any injection | Within 30 minutes of any/each injections
  Number of participants experiencing immediate AEs
Presence of solicited injection site reactions through 7 days after each/any injection | Through 7 days after each/any injections
  Number of participants experiencing solicited injection site reactions
Presence of solicited systemic site reactions through 7 days after each/any injection | Through 7 days after each/any injections
  Number of participants experiencing solicited systemic site reactions
Presence of unsolicited AEs through 21 days after the first injection and through 28 days after the second injection | Through 21 days after the first injection and through 28 days after the second injection
  Number of participants experiencing unsolicited AEs
Presence of medically attended adverse events (MAAEs) through 180 days after the last injection | Through 180 days after the last injection
  Number of participants experiencing MAAEs
Presence of adverse events of special interest (AESIs) throughout the study | Throughout the study, approximately 13 months
  Number of participants experiencing AESIs
Presence of serious adverse events (SAEs) throughout the study | Throughout the study, approximately 13 months
  Number of participants experiencing SAEs
Presence of out-of-range biological test results (including shift from baseline values) through a maximum of 8 days after each injection | Through a maximum of 8 days after each injection
  Number of participants with out-of-range biological test results

SECONDARY OUTCOMES:
Antibody titers measured by Hemagglutination Inhibition (HAI) Assay | At Day 01, Day 22, Day 43, Day 112, and Day 202
  Antibody titers are expressed as geometric mean titers (GMTs)
Individual HAI titer ratio | At Day 22/Day 01, Day 43/Day 01, Day 112/Day 01, and Day 202/Day 01
≥ 4-fold increase in HAI titer [1/dilution]) | At Day 22 or Day 43
HAI titer ≥ 10 [1/dilution] | At day 01
HAI titer ≥ 40 [1/dilution] | At Day 01, Day 22, Day 43, Day 112, and Day 202
Detectable HAI titer ≥ 10 [1/dilution] | At Day 01, Day 22, Day 43, Day 112, and Day 202
Antibody titers measured by Seroneutralization (SN) test | At Day 01, Day 22, Day 43, Day 112, and Day 202
  Antibody titers are expressed as GMTs
Individual SN titer ratio | Day 22/Day 01, Day 43/Day 01, Day 112/Day 01, and Day 202/Day 01
SN titer ≥ 20 (1/dilution) | At Day 01, Day 22, Day 43, Day 112, and Day 202
SN titer ≥ 40 (1/dilution) | At Day 01, Day 22, Day 43, Day 112, and Day 202
SN titer ≥ 80 (1/dilution) | At Day 01, Day 22, Day 43, Day 112, and Day 202
Detectable SN titer ≥ 10 (1/dilution) | At Day 01, Day 22, Day 43, Day 112, and Day 202
2-fold rise in SN titer | At Day 22 and Day 43
4-fold rise in SN titer | At Day 22 and Day 43

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Velocity Clinical Research - San Diego- Site Number : 8400013, La Mesa, California
  - Accel Research Sites Network - DeLand Clinical Research Unit- Site Number : 8400002, DeLand, Florida
  - ARSN-Lakeland CRU- Site Number : 8400006, Lakeland, Florida
  - Accel Research Sites - St. Petersburg- Site Number : 8400004, Largo, Florida
  - Atlanta Clinical Research Center- Site Number : 8400007, Atlanta, Georgia
  - Accel Research Site - NeuroStudies.net, LLC - ERN - PPDS- Site Number : 8400003, Decatur, Georgia
  - QUEST Research Institute- Site Number : 8400014, Bingham Farms, Michigan
  - Velocity Clinical Research - Norfolk- Site Number : 8400015, Norfolk, Nebraska
  - Velocity Clinical Research - Omaha- Site Number : 8400012, Omaha, Nebraska
  - Velocity Clinical Research - Springdale- Site Number : 8400010, Cincinnati, Ohio
  - Coastal Carolina Research Center - North Charleston- Site Number : 8400001, North Charleston, South Carolina
  - Olympus Clinical Research - Sugar Land- Site Number : 8400009, Sugar Land, Texas
  - Velocity Clinical Research, Salt Lake City- Site Number : 8400011, West Jordan, Utah
  - Charlottesville Medical Research- Site Number : 8400005, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VBS00001 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26358&tenant=MT_SNY_9011